CLINICAL TRIAL: NCT04648761
Title: OPTIMAL - Individualized Titration of Biologics in Severe Asthma
Brief Title: Individualized Titration of Biologics in Severe Asthma
Acronym: OPTIMAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Celeste Porsbjerg, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMAL
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: One group will have their biological treatment titrated via the OPTIMAL algorithm and a control group will continue their biological treatment unchanged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OPTIMAL group (Experimental): This group will have their anti IL 5 biologics titrated by OPTIMAL algorithm
  Interventions: Biological: OPTIMAL algorithm
- Control group (No Intervention): This group will continue their treatment with anti IL 5 biologics unchanged

INTERVENTIONS:
Biological: OPTIMAL algorithm — The OPTIMAL algorithm titrates anti IL 5 treatment by addjusting the intervals between injections by FEV1, blood eosinophils and exacerbations.
  Arms: OPTIMAL group

SUMMARY:
OPTIMAL is a non-inferiority, open label randomized clinical trial thats investigates a titration algorithm for anti IL 5 biologics in severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* Age > 18 years
* Correct asthma diagnosis as judged by (sub)-investigator
* Treatment with anti-IL5/IL5r for 12 months or longer
* Treatment with the same biologic drug in the last 12 months
* No exacerbations requiring OCS in the last 12 months
* Blood eosinophils < 0.30 in the last 12 months
* No daily OCS for more than 3 days in the last 12 months with asthma as indication
* Correct inhalation technique for using regular inhalers
* Acceptable adherence to ICS (according to FMK as judged by (sub)-investigator)

Exclusion Criteria:

* - Pregnant or breastfeeding females
* Lack of effective contraception in women of childbearing potential who are sexually active with a non-sterilized male partner. Women of childbearing potential are defined as those who are not surgically sterile (e.g. bilateral tubal ligation, bilateral oophorectomy, complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Effective contraception is defined as intrauterine device (hormonal or non-hormonal), sexual abstinence, bilateral tubal occlusion, combined (estrogen and progesterone) hormonal contraception (oral, intravaginal and transdermal) and progesterone-only hormonal contraception (oral, injectable and implantable).
* Previous medical history or evidence of an uncontrolled intercurrent illness such as but not limited to (e.g. Autoimmune disease, immunodeficiency, immunosuppression, malignant neoplastic conditions with current relevance) that in the opinion of the investigator may compromise the safety of the subject in the study or interfere with evaluation of the algorithm or reduce the subject's ability to participate in the study. Subjects with well-controlled comorbid disease (eg, hypertension, hyperlipidaemia, gastroesophageal reflux disease) on a stable treatment regimen for 15 days prior to inclusion are eligible.
* Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the algorithm or interpretation of subject safety or study results (eg. chronic obstructive pulmonary disease, cystic fibrosis, pulmonary fibrosis, bronchiectasis, allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis polyangitiis, alpha-1-antitrypsin deficiency, Wegeners granulomatosis, Sarcoidosis).
* Any clinically relevant abnormal findings in haematology or clinical chemistry (laboratory results from Visit 0), physical examination, vital signs during the screening, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of chronic alcohol- or drug abuse 12 months prior to inclusion
* Concurrent enrolment in another clinical study involving an investigational treatment.
* Use of immunosuppressive medication (eg, methotrexate, troleandomycin, oral gold, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroids or any experimental anti-inflammatory therapy) within 3 months prior to inclusion and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of proportions of patients with exacerbations aften one year in each group | one year

SECONDARY OUTCOMES:
Proportion of patients on reduced dose of biologics at the end of trial | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Research Unit, Med. Clinic I, Bispebjerg Hospital, Bispebjerg Bakke 23, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No